CLINICAL TRIAL: NCT03595501
Title: Analytical and Clinical Performance Testing Plan
Status: Completed | Type: Observational
Sponsor: Sight Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: PR00014
Record Dates: First submitted 2018-05-28; First posted 2018-07-23 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Hematology; Hematologic Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Hematology Analyzer - OLO: The investigational device is a quantitative multi-parameter automated hematology analyzer intended for in vitro diagnostic use in screening capillary or venous whole blood samples.
  Interventions: Device: Hematology Analyzer - OLO
- Hematology Analyzer - Predicate: The predicate device is a quantitative multi-parameter automated hematology analyzer intended for in vitro diagnostic use in screening patient populations found in clinical and reference laboratories.
  Interventions: Device: Hematology Analyzer - Predicate

INTERVENTIONS:
Device: Hematology Analyzer - OLO — Complete blood counts from OLO will be determined from analysis of whole blood samples
  Groups: Hematology Analyzer - OLO
Device: Hematology Analyzer - Predicate — Complete blood counts from Predicate will be determined from analysis of whole blood samples
  Groups: Hematology Analyzer - Predicate

SUMMARY:
Clinical and analytical tests will be performed based on risk assessment and system specifications to verify that the performance of the investigational device is in accordance with its specifications.

DETAILED DESCRIPTION:
Comparison and precision studies will be conducted in up to 5 clinical sites in Israel and the US, and include:

* Precision
* Sample Matrix Comparison
* Method comparison study and flagging analysis
* Reference interval range

ELIGIBILITY:
Inclusion Criteria:

For Residual Samples:

* Specimen obtained by venipuncture or finger prick and collected into tubes normally used by the site
* Patient is at least 3 months of age
* Samples within 8 hours from phlebotomy

For Prospectively collected samples:

* Subject is at least 22 years of age
* Non-diseased individuals or, for specific studies, individuals with blood count ranges to cover indicated medical decision points and ranges
* Samples within 8 hours from phlebotomy

Exclusion Criteria:

Exclusion criteria post blood draw and pre sample scan - For whole blood samples:

* Visibly hemolyzed or clotted specimens
* Specimens with insufficient blood volume to complete the procedure
* Samples older than eight hours

Exclusion criteria post sample scan:

* Instrument failure or sample rejected by the instrument due to system error or sample mishandling
* The daily quality control sample measurements indicate that the assay run is outside the specifications for the instrument
* Operator related error documented in the study records
* Failure to adhere to study specifics or protocols

Min Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adult and pediatric patients with normal (healthy) or abnormal blood counts (known clinical condition)
Sampling Method: Non-Probability Sample
Enrollment: 679 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-08-25 (Actual)

PRIMARY OUTCOMES:
Reproducibility of CBC parameters provided by the OLO device | 3 months
  Reproducibility studies will be conducted using 3 levels of commercial control materials (low, normal and high) to measure all CBC reported parameters. Control material will be run on two instruments at each site. Standard deviation (SD) and coefficient of variation (CV) will be calculated for each measurand for: (1) Between lots/sites; (2) Between instruments; (3) Between days; (4)Between operators/runs; (5) within-run and (6) total variability
Repeatability of CBC parameters provided by the OLO device | 3 months
  Performance of the OLO device will be measured through repeatability of 20 replicates for 11 residual samples on each site. Samples collected for this study will include 4 within lab reference range, 3 around lower medical decision levels for HGB, PLT and WBC, and 4 around the upper range for RBC, HGB, WBC and PLT to cover all pathological levels and medical decision points. Standard deviation (SD) and coefficient of variation (CV) will be computed for each measurand per sample by site.
Sample Matrix Comparison | 3 months
  Paird capillary and venous whole blood samples will be collected. The samples will be analyzed in duplicate on the Sight OLO device. Analysis will include Passing-Bablok Regression analysis per parameter (Bland Altman plots, slope, intercept, with 95% confidence intervals, correlation coefficient, and % bias), between: The average of venous whole blood samples scans and average of capillary whole blood sample scans from the same individual on the Sight OLO device
Method Comparison | 3 months
  Evaluate the performance of the OLO device in comparison to values achieved with the predicate. Analysis will include Regression parameters (slope, intercept with 95% CI) between measurement of Sight OLO and measurement on predicate (Correlation coefficient, Bland Altman plots and overall % bias between predicate and Sight OLO device including % bias at medical decision points).
Reference Interval Range | 3 months
  Establish adult venous and fingerprick reference intervals for the OLO device. The non-parametric method will be used to calculate the lower and upper limits of the reference range.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Eldad Hod, Dr, Principal Investigator — Colombia University
Locations (1):
- Columbia University, New York, New York, United States